CLINICAL TRIAL: NCT05117918
Title: A Prospective Study Evaluating the Feasibility of Telemedicine Use in the Overactive Bladder Clinical Care Pathway: a Non-inferiority Study Assessing Patient Satisfaction and Progression to Third Line Overactive Bladder Therapies
Brief Title: Overactive Bladder Telemedicine Non-inferiority Trial
Acronym: OAB Telemed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Victor W. Nitti, MD, Professor of Urology, Chief, Division of Female Pelvic Medicine and Reconstructive Surgery, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-000458
Record Dates: First submitted 2021-08-18; First posted 2021-11-11 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Telemedicine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional In-Person Clinic Visit Arm (Placebo Comparator): Patients will receive overactive bladder (OAB) treatment as described in the Society for Urodynamics and Female Pelvic Medicine and Urogenital Reconstruction (SUFU) OAB clinical care pathway. These patients will have all visits in-person
  Interventions: Other: SUFU Clinical Care Pathway for Overactive Bladder
- Telemedicine Arm (Experimental): Patients will receive OAB treatment as described in the SUFU OAB clinical care pathway but all visits will be performed via telemedicine
  Interventions: Other: SUFU Clinical Care Pathway for Overactive Bladder; Other: Telemedicine

INTERVENTIONS:
Other: SUFU Clinical Care Pathway for Overactive Bladder — Treatment of OAB via the SUFU clinical care pathway
Other: Telemedicine — Delivery of care via telemedicine
  Arms: Telemedicine Arm

SUMMARY:
In this study, the investigators aim to validate the telemedicine paradigm as a feasible alternative to traditional in-person clinic visits for the management of overactive bladder (OAB).

DETAILED DESCRIPTION:
This is a single-center, prospective randomized controlled trial. The study population will consist of two primary cohorts stratified based on the method of follow-up, either traditional in-person clinic visit or telemedicine appointment. The primary outcome will be satisfaction with OAB treatment. Secondary endpoints include rate of progression to third line therapies, changes in OAB symptom scores, safety, and cost. This non-inferiority trial is designed to provide an alternative option for care delivery that may result in improved patient satisfaction and compliance, and decreased cost, time, and travel burden for patients.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic overactive bladder diagnosis, both OAB wet and OAB dry

Exclusion Criteria:

* Active Urinary Tract Infection (UTI)
* Stage 3 or 4 prolapse
* Underlying neurologic condition contributing to OAB
* Use of catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | 1 year
  Treatment Satisfaction Visual Analogue Scale (TS-VAS), scale scored from 0 - 100 with 100 indicating highest satisfaction

SECONDARY OUTCOMES:
PGII | 1 year
  Patient Global impression of improvement (PGII), minimum of 0, maximum of 6 with 0 indicating the patient is most improved
Incidence of Treatment-emergent adverse events (safety and tolerability) | 1 year
  Adverse events related to treatment requiring emergency room visits, urgent care visits, hospital admissions
Accumulated cost of visit to patient (Cost) | 1 year
  Cost of parking, travel, and other visit-associated expenses to patient
Accumulated time of visit for patient (Time) | 1 year
  Time of travel to visit, time of visit, wait time of visit
Overactive Bladder Symptoms | 1 year
  Overactive Bladder Questionnaire Short-Form (OAB-q SF), scale from 6-36 with 36 indicating the most severe OAB symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States